CLINICAL TRIAL: NCT05980988
Title: Efficacy and Safety of Probiotic BLa80 in Modulating Bowel Habits in Subjects With Chronic Constipation
Brief Title: Effectiveness and Safety of Probiotic in Regulating Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Collaborators: Methodex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK2023003
Record Dates: First submitted 2023-07-28; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Chronic Constipation
Keywords: Probiotics；Chronic constipation
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double（Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): 2B CFU/capsule/day BLa80, before meals； Storage: Store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Probiotic
- placebo (Placebo Comparator): Maltodextrin, one capsule/day, before meals； Storage: Store in a cool, dry place without exposure to the sun.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of this study had last 84 days, and each patient will make 4 visits (d1, d28, d56, d84).
  Arms: Probiotic group
Dietary Supplement: Placebo — Placebo
  Arms: placebo

SUMMARY:
To evaluate the effectiveness and safety of the use of probiotics as food supplements in regulating the intestinal habit of subjects with chronic constipation, in comparison with placebo.

ELIGIBILITY:
Inclusion Criteria:

Patients with chronic constipation (duration more than 3 months with less than three bowel movements per week and/or Bristol Scale 1 and 2).

Exclusion Criteria:

1. Diabetic patients.
2. Pregnant patients.
3. Breastfeeding patients.
4. Patients requiring antibiotic treatment.
5. Patients requiring treatment with tricyclic antidepressants, antiepileptics, antihistamines, antiparkinsonians, antipsychotics, antispasmodics, verapamil, monoamine oxidase inhibitors, opiates, sympathomimetics, antacids (with aluminum and calcium), antidiarrheals and nonsteroidal anti-inflammatory drugs.
6. Patients who change the type of diet during the study.
7. Patients with allergy or intolerance to any of the ingredients in the formulation of the product under study.
8. Subjects with a history of pharmacological, alcoholic, or other substance abuse, or other factors that limit their ability to cooperate during the study.
9. Excessive alcohol consumption (>3 glasses of wine or beer/day).
10. Subjects whose condition does not make them eligible for the study, according to the researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
changes in fecal state | 84 days
  use Bristol Scale to record the type of fecal state

CONTACTS AND LOCATIONS:
Overall Officials: METHODEX SL, Study Chair — Methodex
Locations (2):
- Spain (2):
  - CAP Can Bou Castelldefels and CAP Corbera de Llobregat, Barcelona
  - Family and Community Medicine CAP Roger, Barcelona

REFERENCES:
- [Derived] Salo E, Roche D, Gomez-Martinez VB, Cruz-Domenech JM, Garcia-Mora LG, Gabernet-Castello C, Freixenet N. Bifidobacterium animalis subsp. lactis BLa80 regulates the intestinal habit in adults with chronic constipation: a multicentre, randomised, double-blind, placebo-controlled study. Benef Microbes. 2024 Sep 5;15(6):679-688. doi: 10.1163/18762891-bja00038. PMID 39244201